CLINICAL TRIAL: NCT06296381
Title: Analysis of Peripheral Muscle Strength Measurement Methods in Healthy Individuals and Critical Patients: A Health Technology Assessment
Brief Title: Normative Values for Peripheral Muscle Strength in Critical Patients and Healthy Individuals
Acronym: HHD-ICU
Status: Recruiting | Type: Observational
Sponsor: University of Pernambuco (Other)
Collaborators: Universidade Federal de Pernambuco (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Shirley Lima Campos, Associate Professor, University of Pernambuco
Other Study IDs: 6.131.540
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Intensive Care Unit; Muscle Strength
Keywords: Healthy Volunteers; Critically ill; Peripheral muscle
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients in the ICU: The ICU sample will comprised patients of both sexes, aged between 18 and 90 years old, able to do volitional tests and without barriers to the assessment of peripheral muscle strength.
- Healthy Participants: The healthy sample will comprised volunteers of both sexes, aged between 18 and 90 years old, able to do volitional tests and without barriers to the assessment of peripheral muscle strength.

SUMMARY:
Muscle strength is an important indicator of overall health and is a factor that has been associated with increased mortality in critical patients. Its measurement must be reliable and reproducible to ensure a quality outcome for clinical applicability. Recently, the use of digital handheld dynamometers in intensive care has gained support; however, analysis becomes challenging due to the absence of standardized reference equations for the Brazilian population. The aim of this study is to develop reference equations for the Brazilian population and define specific cutoff points for men, women, healthy individuals, and critical patients.

DETAILED DESCRIPTION:
For this 3-year observational study, the population will consist of adult and elderly individuals of both sexes; for the healthy sample, patients without barriers to the assessment of peripheral muscle strength will meet the inclusion criteria, specifically, areas with wounds/dressings, burns, segments with fractures, or immobilization devices, while, for the critical patient population, the sample will comprise patients who are hospitalized in the Intensive Care Unit (ICU).

In the case of assessing healthy participants, an evaluation of the musculoskeletal system will be conducted to measure muscle strength (handgrip dynamometry and peripheral hand held muscle dynamometry). Regarding critical patients, if the participant meets the criteria, the evaluation protocol will be carried out, which includes peripheral muscle strength assessment (Medical Research Council scale, Hand Dynamometer, and the Hand-Held Dynamometer) and the patient's mobility status (ICU Mobility Scale).

Daily screening will take place in the ICU, with eligibility assessed during the screening process. If eligible, secondary data related to the critical condition will be extracted from the participant's medical records, including anthropometric data, sociodemographic information, neurological and cardiovascular assessments, current medications, and laboratory test results. The participant's hemodynamic and respiratory stability will be monitored using a multiparameter monitor, recording data such as blood pressure, heart rate, peripheral saturation, and respiratory rate. A cardiorespiratory and clinical safety checklist will also be completed prior to conducting tests for all patients, regardless of whether they are using mechanical ventilation. The instruments used for assessment the muscle strength are the Digital Hand Dynamometer (Saehan Corporation®, DHD-1) and the Hand Held Dynamometer (HOGGAN SCIENTIFIC LLC, microFET2).

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals of both sexes
* Patients and volunteers aged between 18 and 90 years old (youth/adults/elderly).
* Patients admitted to the ICU.
* No recent muscle injuries of both limbs for a past 6-months.

Exclusion Criteria:

Patients and volunteers < 20 years and > 90 years

Healthy individuals

* Unable to follow command completely
* Severe osteoporosis or neuromuscular disease leading to decreased muscle strength
* Presence of opened or infectious wound
* Presence of pain in evaluating muscle groups

Patients in ICU

* Unable to follow command completely
* Acute stroke
* Hip fracture, unstable cervical spine or pathological fracture
* Recent surgery involving the upper airways, chest, abdomen, or limbs
* Presence of opened or infectious wound
* Presence of pain in evaluating muscle groups

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population comprised adult and elderly individuals of both sexes able to do volitional tests. For the healthy sample, volunteers without barriers to the assessment of peripheral muscle strength will meet the inclusion criteria while, for the critical patient population, the sample will include individuals hospitalized in the Intensive Care Unit (ICU) who also do not have barriers to the assessment.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Peripheral muscle strength measured by hand held dynamometer | Day 1
  Strength of the muscles of the upper and lower limbs using a digital hand held dynamometer in healthy individuals and critical patients.
Peripheral muscle strength measured by Medical Research Council score | Day 1
  Global muscle strength using the Medical Research Council-sum score (MRC score) in healthy individuals and critical patients. The MRC score is obtained by evaluating muscle groups in the upper and lower extremities (wrist extensors, elbow flexors, abductors of the shoulder, dorsal ankle flexors, knee extensors, and hip flexors). For each muscle group will be assigned a score between 0 and 5, and the total score can vary between 0 (worse outcome) up to 60 points (the better outcome).

SECONDARY OUTCOMES:
Peripheral muscle strength measured by hand grip dynamometer | Day 1
  Peripheral muscle strength assessed bilaterally through digital handgrip dynamometry in healthy individuals and critical patients.
Level of activity in ICU at the moment | Day 1
  The ICU Mobility Scale is a tool used to assess mobility milestones in critically ill patients, categorizing them on a scale from 0 to 10 as follows: (0) no mobility (lying in bed), (1) sitting in bed (performing exercises), (2) passively moved to a chair (without standing), (3) sitting at the edge of the bed, (4) standing, (5) transferring from bed to chair, (6) marching in place (at the bedside), (7) walking with assistance from two or more people, (8) walking with assistance from one person, (9) walking independently with a gait aid, and (10) walking independently without a gait aid. The scale ranges from a minimum of 0 to a maximum of 10, with higher scores indicating better functional outcomes.
Level of frailty in healthy older adults by the Multidimensional Assessment of Older People (AMPI-AB) | Day 1
  The AMPI-AB is composed of 17 questions based on well-known and validated scores used to detect relevant geriatric problems, such as lack of social support, multimorbidity, polypharmacy, cognitive and sensory impairment, physical limitations, depression, falls, functional dependence, weight loss and poor oral health. The total score can vary between 0 (the best outcome) up to 21 (the worst outcome) and classifies older adults in low, intermediate or high complexity of care.
Level of frailty in ICU older adults by the Clinical Frailty Scale (CFS) | Day 1
  The Clinical Frailty Scale (CFS) is a well-validated tool developed to quantify the degree of frailty and disability in older adults. It is based on clinical judgment and provides a global measure of vulnerability to adverse health outcomes. The scale ranges from 1 (very fit, the best outcome) to 9 (terminally ill, the worst outcome), with each incremental score reflecting a greater degree of frailty, functional dependence, and health decline. The CFS is supported by a visual chart that guides clinicians in the classification of frailty levels.
Adverse Events | Day 1
  An adverse event is defined as any unfavorable or unintended medical sign, symptom, or condition that arises during or after the peripheral muscle strength assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Vinicius Porfirio, Principal Investigator — University of Pernambuco; Shirley Campos, Study Chair — University of Pernambuco
Locations (4):
- Brazil (4):
  - Complexo Hospitalar Unimed Recife - CHUR, Recife, Brazil
  - Federal University of Pernambuco (UFPE), Recife, Pernambuco
  - Hospital Otávio de Freitas, Recife, Pernambuco
  - Hospital Nossa Senhora das Graças, Recife, Pernambuco

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lumbroso L, Doz F, Urbieta M, Levy C, Bours D, Asselain B, Vedrenne J, Zucker JM, Desjardins L. Chemothermotherapy in the management of retinoblastoma. Ophthalmology. 2002 Jun;109(6):1130-6. doi: 10.1016/s0161-6420(02)01053-9. PMID 12045055
- [Background] Teale JD. The diagnostic application of serum growth hormone, insulin-like growth factor (IGF), and IGF binding protein measurements. J Int Fed Clin Chem. 1995 Nov;6(5):164-8. PMID 10155148
- [Background] Saraiva MD, Venys AL, Abdalla FLP, Fernandes MS, Pisoli PH, Sousa DMDRV, Bianconi BL, Henrique EA, Garcia VSS, Maia LHM, Suzuki GS, Serrano PG, Hiratsuka M, Szlejf C, Jacob-Filho W, Paschoal SMP. AMPI-AB validity and reliability: a multidimensional tool in resource-limited primary care settings. BMC Geriatr. 2020 Mar 30;20(1):124. doi: 10.1186/s12877-020-01508-9. PMID 32228469
- [Background] Samosawala NR, Vaishali K, Kalyana BC. Measurement of muscle strength with handheld dynamometer in Intensive Care Unit. Indian J Crit Care Med. 2016 Jan;20(1):21-6. doi: 10.4103/0972-5229.173683. PMID 26955213
- [Background] Stark T, Walker B, Phillips JK, Fejer R, Beck R. Hand-held dynamometry correlation with the gold standard isokinetic dynamometry: a systematic review. PM R. 2011 May;3(5):472-9. doi: 10.1016/j.pmrj.2010.10.025. PMID 21570036
- [Background] Nunez-Cortes R, Cruz BDP, Gallardo-Gomez D, Calatayud J, Cruz-Montecinos C, Lopez-Gil JF, Lopez-Bueno R. Handgrip strength measurement protocols for all-cause and cause-specific mortality outcomes in more than 3 million participants: A systematic review and meta-regression analysis. Clin Nutr. 2022 Nov;41(11):2473-2489. doi: 10.1016/j.clnu.2022.09.006. Epub 2022 Sep 16. PMID 36215867